CLINICAL TRIAL: NCT02237534
Title: Lanthanum Carbonate Versus Calcium Carbonate for Vascular Abnormalities in Patients With Chronic Kidney Disease and Hyperphosphatemia
Brief Title: Lanthanum Versus Calcium Carbonate for Vascular Abnormalities in Patients With CKD and Hyperphosphatemia
Acronym: LAVALIER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Osaka University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Takayuki Hamano, Endowed chair, Osaka University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKDR-002
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Renal Insufficiency, Chronic; Hyperphosphatemia; Bone Diseases, Metabolic
Keywords: Lanthanum; Calcium Carbonate; Vascular Calcification
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia; Bone Diseases, Metabolic; Vascular Calcification | interventions — lanthanum carbonate; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium carbonate (Active Comparator): Start at a dose of 1,500 mg/day, and adjust it to lower serum phosphate concentration <4.5 mg/dL. Maximum dose is 3,000 mg/day.
  Interventions: Drug: Calcium Carbonate
- Lanthanum carbonate (Experimental): Start at a dose of 750 mg/day, and adjust it to lower serum phosphate concentration <4.5 mg/dL. Maximum dose is 1,500 mg/day. For patients with calcium carbonate at inclusion, calcium carbonate will be replaced with lanthanum carbonate of 750 mg/day.
  Interventions: Drug: Lanthanum carbonate

INTERVENTIONS:
Drug: Lanthanum carbonate
  Other Names: FOSRENOL®
  Arms: Lanthanum carbonate
Drug: Calcium Carbonate
  Arms: Calcium carbonate

SUMMARY:
The purpose of this study is to compare the effect of lanthanum carbonate and calcium carbonate on the progression of coronary calcification and vascular endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Hyperphosphatemia (For patients without calcium carbonate, ≥4.5 mg/dL) (For patients with calcium carbonate, ≥4.0 mg/dL)
* With written informed consent

Exclusion Criteria:

* History of cardiac surgery
* With coronary artery stent
* Polycystic kidney disease
* Hypothyroidism
* On treatment with lanthanum carbonate
* History of admission within 3 months
* History of ileus
* Severe liver dysfunction
* Severe gastrointestinal dysfunction
* Allergy to lanthanum carbonate or calcium carbonate
* Pregnant or breastfeeding women
* Judged as ineligible by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Coronary artery calcification score | 1 year

SECONDARY OUTCOMES:
Endothelial function | 3 months
  Measured by EndoPAT™ (Itamar Medical Ltd.)
Serum bone metabolic markers | 3 months
  Bone specific alkaline phosphatase (BAP) and Tartrate-resistant acid phosphatase 5b (TRACP5b)
Serum bone metabolic markers | 1 year
  Bone specific alkaline phosphatase (BAP) and Tartrate-resistant acid phosphatase 5b (TRACP5b)
Serum concentrations of calcium, phosphate, intact parathyroid hormone, 25-hydroxyvitamin D, and 1,25-dihydroxyvitamin D over time | Up to 1 year
Estimated glomerular filtration rate over time | Up to 1 year
Bone mineral density | 1 year
Serum osteoprotegerin concentration | 3 month
Serum osteoprotegerin concentration | 1 year
Urinary alpha-Klotho to creatinine ratio | 3 months
Urinary alpha-Klotho to creatinine ratio | 1 year
Urinary liver-type fatty acid binding protein (L-FABP) to creatinine ratio | 3 months
Urinary liver-type fatty acid binding protein (L-FABP) to creatinine ratio | 1 year
End-stage renal disease requiring renal replacement therapy | Up to 1 year
Cardiovascular event requiring hospitalization | Up to 1 year
  Acute myocardial infarction, angina pectoris, congestive heart failure, stroke, and peripheral vascular disease
Death | Up to 1 year

OTHER OUTCOMES:
Micro RNA array | 1 year
Hypercalcemia | Up to 1 year
  Corrected serum calcium concentration ≥11.0 mg/dL
Hypocalcemia | Up to 1 year
  Corrected serum calcium concentration <8.5 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Takayuki Hamano, MD, PhD, Study Chair — Department of Comprehensive Kidney Disease Research, Osaka University Graduate School of Medicine
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan